CLINICAL TRIAL: NCT02283593
Title: Self-help Internet-based Relapse Prevention for Problematic Alcohol Use: A Naturalistic Study Among Internet Help-seekers
Brief Title: Self-help Internet-based Relapse Prevention for Problematic Alcohol Use
Acronym: eChangeNAT
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anne H Berman, Associate Professor, Karolinska Institutet
Other Study IDs: 2013/686-31/5; KI 2-1341/2014 (Other: Karolinska Institutet, Personal data act registrar)
Record Dates: First submitted 2014-11-02; First posted 2014-11-05 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Problematic Alcohol Use

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: eChange.se — 7 modules: 1. Making a decisional balance 2. Setting a goal for alcohol consumption 3. Learning self control skills 4. Identifying risk situations 5. Dealing with urges 6. Dealing with emotions and with social pressure 7. Developing a crisis plan
  Other Names: SO (Self-help online, see Blankers et al., 2011)

SUMMARY:
The purpose of this study is to observe and evaluate the use of a relapse prevention program over time among internet help-seekers. Participants are recruited via a nationally known portal for assisting anonymous individuals with changing their problematic alcohol use in a healthier direction (alkoholhjalpen.se). The intervention offered lasts 10 weeks and includes 7 relapse prevention modules, with a three-week pause between the 6th and 7th modules. Baseline data are collected regarding substance use and psychosocial health and follow-up takes place 10 weeks after recruitment. The study is observational.

ELIGIBILITY:
Inclusion Criteria:

* AUDIT >5 points for women
* AUDIT >7 points for men

Exclusion Criteria:

* AUDIT <6 points for women
* AUDIT <8 points for men

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Internet help-seekers with problematic alcohol use.
Sampling Method: Non-Probability Sample
Enrollment: 4165 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Timeline Follow Back (TLFB) | 10 weeks
  Quantity/frequency measure of alcohol consumption
The Alcohol Use Disorders Identification Test (AUDIT) | 10 weeks
  3 consumption questions and 7 problem-related questions regarding alcohol consumption

SECONDARY OUTCOMES:
The Drug Use Disorders Identification Test (DUDIT) | 10 weeks
  3 consumption questions and 7 problem-related questions regarding drug consumption
The Hospital Anxiety and Depression Scale (HADS) | 10 weeks
  14 questions, 7 on anxiety symptoms and 7 on depression symptoms
The Readiness to Change Questionnaire (RTCQ) | 10 weeks
  12 questions rated from -2 to +2 and divided into 3 dimensions: precontemplation, contemplation and action
The Readiness Ruler | 10 weeks
  Scores between 0 and 100. In this study, "I am not ready to change my drinking habits" and "I am very much ready to change my drinking habits".
The World Health Quality of Life - shorter version (WHOQOL - BREF) | 10 weeks
  26 questions measuring four domains of quality of life: physical, psychological, social and environment.
EQ-5D-5L | 10 weeks
  5 questions on the following dimensions: mobility, self-care, usual activity, pain/discomfort and anxiety/discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Department of Clinical Neuroscience, Stockholm, Sweden

REFERENCES:
- [Background] Sinadinovic K, Wennberg P, Johansson M, Berman AH. Targeting individuals with problematic alcohol use via Web-based cognitive-behavioral self-help modules, personalized screening feedback or assessment only: a randomized controlled trial. Eur Addict Res. 2014;20(6):305-18. doi: 10.1159/000362406. Epub 2014 Oct 4. PMID 25300885